CLINICAL TRIAL: NCT02481232
Title: A Single-center, Open Trials to Evaluate the Safety of Freeze-dried Group ACYW135 Meningococcal Conjugate Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCV4-001
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Meningococcal Meningitis
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- freeze-dried group ACYW135 MCV 4μg (Experimental): 4μg group: vaccines serial number is A0001-A0100（18-55 years-old group A0001-A0020，7-17 years-old group A0021-A0040，1-6 years-old group A0041-A0060，7-10 months-old group A0061-A0080，2 months-old group A0081-A0100）
  Interventions: Biological: freeze-dried group ACYW135 MCV
- freeze-dried group ACYW135 MCV 8μg (Experimental): 8μg group: vaccines serial number is B0001-B0100（18-55 years-old group B0001-B0020，7-17 years-old group B0021-B0040，1-6 years-old group B0041-B0060，7-10 months-old group B0061-B0080，2 months-old group B0081-B0100）
  Interventions: Biological: freeze-dried group ACYW135 MCV

INTERVENTIONS:
Biological: freeze-dried group ACYW135 MCV — Group A, C, Y and W135 Meningococcal conjugate vaccine is suitable for immune prevention of epidemic cerebrospinal meningitis more than 2 months of age population

SUMMARY:
Safety Evaluation of freeze-dried Group ACYW135 Meningococcal conjugate vaccine in healthy people above 2-months-old

DETAILED DESCRIPTION:
There are five different age groups(18~55 years/7~17 years/1~6 years/7~10 months/2 months),each group has 40 people and divided into two subgroups. Each subgroup will inject different vaccine(MCV4 4μg,MCV4 8μg).For 7~10 months&2 months age groups,there are 2&3 injection seperately. Each injection interval is 1 months.

After 7 days observation of 1 dose immunization in Group 18-55 years old adults, if there are no serious adverse events associated with vaccines, or severe adverse reactions rate is less than 10%, 7 to 17 years old and 1 to 6 years old age groups will continue to inoculate in order. After the first dose of 7~10 months group and evaluating safety, 2 months group immunized the first dose. All participants completed the immune procedure, then observed the safety to 30 days after whole immunization.

Data collection: Subjects completed diary card, the researchers collected original data and fill out the case report form for data entry and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants unimmunized Group A&C meningococcal conjugate vaccine or Group A meningococcal polysaccharide vaccine which is above 2~11 months-old, and healthy toddler more than 1-year-old without booster immunization.
* The guardian or himself informed consent, and signed the informed consent form;
* The guardian and family agreed to abide by the requirements of clinical trial scheme;
* Participants has no history of immunoglobulin vaccination in the last 2 months / 2 months-old infants has no history of immunoglobulin vaccination after born, there is no history of other live vaccine inoculation before vaccination in 14 days, within 7 days without other inactivated vaccine immunization history;
* the axillary temperature < 37.1 ℃;
* 2-months-old group in the age of 61-90 days;
* 7-months-old group in the age of 211-300 days;
* 1-year-old group in age of one full year of life.

Exclusion Criteria:

* Have allergies, convulsions, seizures, encephalopathy and psychiatric history or family history;
* Neomycin, streptomycin and polymyxin B allergies;
* With immunodeficiency, immunosuppressant therapy;
* History of meningitis;
* Women in lactation or pregnant;
* Acute febrile diseases and infectious diseases;
* History of labor abnormalities, choking rescue, congenital malformations, developmental disorders or serious chronic disease patients;
* Had a severe allergic reaction of vaccination in the past;
* Took oral steroids more than 14 days in last month;
* Had high fever (axillary temperature≥38.0℃ or higher)in the past three days;
* Prepare to attend or is in any other drug clinical study;
* Meningococcal vaccine contraindications and any situation which researchers think that may affect test evaluation.

Ages: 2 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
systemic and local reactions 30 days after full-course vaccination | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei CDC, Wuhan, Hubei, China